CLINICAL TRIAL: NCT02208011
Title: A Comparison of Rapid Immunoassays for the Detection of Ruptured Membranes
Status: Completed | Type: Observational
Sponsor: Louisiana State University, Baton Rouge (Other)
Collaborators: Woman's Hospital, Louisiana (Other); Clinical Innovations, LLC (Industry); Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Iro Igbinosa, M.D., Louisiana State University, Baton Rouge
Other Study IDs: L8608-W13010
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Evidence of Ruptured Membranes in Women Greater Than 15 Weekd

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Specific objectives include analysis of performance of ROM Plus® in diagnosing ROM, as compared to Amnisure® and the conventional clinical assessment confirmed by a thorough chart review after delivery.

Inclusion Criteria:

* English speaking
* pregnant woman >15 weeks gestation undergoing an exam for ruptured membranes

Exclusion Criteria:

* Known placental previa
* Active vaginal bleeding

ELIGIBILITY:
Inclusion Criteria:

* complaint of ruptured membranes
* IUP > 15 weeks gestation
* English speaking, over the age of 18yrs old

Exclusion Criteria:

* active bleeding
* placenta previa

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant woman presenting to Woman's Hospital, LSU Baton Rouge Clinic with ruptured membranes.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
evidence of ruptured membranes | up to delivery of infant

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Igbinosa I, Moore FA 3rd, Johnson C, Block JE. Comparison of rapid immunoassays for rupture of fetal membranes. BMC Pregnancy Childbirth. 2017 Apr 26;17(1):128. doi: 10.1186/s12884-017-1311-y. PMID 28446135